CLINICAL TRIAL: NCT05029687
Title: A Youth-Led Digital Education Intervention to Improve Blood Pressure for Hypertensive Adults Who Present to the Emergency Department
Brief Title: Youth-Led Intervention to Improve Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Sara Heinert, PhD, MPH, Assistant Professor, Department of Emergency Medicine, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2021000126; UL1TR003017 (NIH)
Record Dates: First submitted 2021-08-19; First posted 2021-08-31 (Actual); Results first posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Hypertension; Adolescent Behavior; Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Hypertension; Adolescent Behavior; Behavior

STUDY DESIGN:
Intervention Model Description: Study transitioned from a randomized controlled trial to a single group study. The total participants enrolled in the trial include all aspects of the study (including qualitative focus groups and interviews).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): The intervention is a youth-led HTN education digital intervention, which will be comprised of a 6-week playlist of one module per week comprising the playlist. Youth will learn from the module and will teach the adult in their dyad about hypertension education in each week's themed module.
  Interventions: Behavioral: Youth-Led Hypertension Education Digital Intervention

INTERVENTIONS:
Behavioral: Youth-Led Hypertension Education Digital Intervention — The intervention is a youth-led HTN education digital intervention, which will be comprised of a 6-week playlist of one module per week comprising the playlist. Youth will learn from the module and will teach the adult in their dyad about hypertension education in each week's themed module.

SUMMARY:
The proposed study will develop, test, and collect implementation data on a youth-led hypertension (HTN) education intervention, which will act as an electronic tool to guide youth through learning and then teaching adults on how to achieve better HTN control. Adults with HTN and youth will be recruited for user-centered design sessions to provide input in the development of a youth-led HTN education digital badge. The investigators will then recruit adult emergency department (ED) patients with uncontrolled HTN (blood pressure (BP) ≥130/80 mm Hg) who know (friend or family member) a youth (14-24 years old) and the youth themselves for a RCT. The adult plus youth dyad will be randomized to either: 1) intervention arm- 6-week youth-led HTN education digital badge at home- or 2) control arm- 6-week youth job readiness digital badge at home. In addition to the primary study outcome of adult BP change 2-months post-intervention, the investigator will collect secondary outcomes of HTN knowledge and youth self-efficacy, as well as implementation metrics of intervention acceptability, feasibility, and fidelity. Due to challenges recruiting youth through adults in the ED, we will be adding a cohort to the study where we will recruit interested youth from New Brunswick Health Sciences Technology High School (NBHSTHS).

Specific aims are:

Aim 1: Create a youth-led HTN education digital badge by means of user-centered design methods and community engagement with adults with HTN and youth to obtain input on the contents of the digital badge prior to implementation.

Aim 1a: The hypertension knowledge assessment being used in the study has not been used before on youth or Spanish-speaking populations, so the investigators will obtain feedback on the assessment from these groups.

Aim 2: Evaluate the effectiveness of a youth-led HTN education digital badge intervention on the primary outcome of mean systolic BP and diastolic BP change in adults with uncontrolled HTN at 2-months post-intervention compared to the control group (for participants recruited from the ED). Additionally, evaluate change in HTN knowledge and youth self-efficacy.

Aim 3: Evaluate the implementation process of the youth-led HTN education digital badge by collecting qualitative and quantitative data on acceptability, feasibility, and fidelity of the intervention by participants.

DETAILED DESCRIPTION:
The proposed study will integrate user-centered design, community engagement, and implementation science, with a randomized controlled trial (RCT), to develop, test, and collect implementation data on a youth-led hypertension (HTN) education digital badge. The badge will act as an electronic tool to guide youth through learning and then teaching adults on how to achieve better HTN control. Adults with HTN and youth will be recruited for user-centered design sessions to provide input in the development of a youth-led HTN education digital badge. The investigators will then recruit adult emergency department (ED) patients with uncontrolled HTN (blood pressure (BP) ≥130/80 mm Hg) who know (friend or family member) a youth (14-24 years old) and the youth themselves for a RCT. The adult plus youth dyad will be randomized to either: 1) intervention arm- 6-week youth-led HTN education digital badge at home- or 2) control arm- 6-week youth job readiness digital badge at home. In addition to the primary study outcome of adult BP change 2-months post-intervention, the investigator will collect secondary outcomes of HTN knowledge and youth self-efficacy, as well as implementation metrics of intervention acceptability, feasibility, and fidelity.

Due to challenges recruiting youth through adults in the ED, we will be adding a cohort to the study. For this new cohort of the study, we will recruit interested youth from New Brunswick Health Sciences Technology High School (NBHSTHS). Students will be asked to pair themselves with an adult (18+) (preference for adult who has been diagnosed with hypertension, but not mandatory) with an existing relationship with the student where it would be feasible to complete an online module together 1 hour per week for 6 weeks. The adult must be fluent in English or Spanish and the student must be able to speak the fluent language of the adult. We will evaluate the youth-led digital hypertension (HTN) education intervention- an electronic tool to guide youth through learning and then teaching and supporting adults on how to control hypertension (for adults with hypertension) and how to avoid it (for adults without hypertension). Outcomes of interest are HTN knowledge, confidence in HTN management, and health behavior changes in participants, which will be obtained through pre- and post- intervention assessments. We will also be exploring outcomes of participant acceptability, feasibility, and fidelity of the intervention.

Specific aims are:

Aim 1: Create a youth-led HTN education digital badge by means of user-centered design methods and community engagement with adults with HTN and youth to obtain input on the contents of the digital badge prior to implementation.

Aim 1a: The hypertension knowledge assessment being used in the study has not been used before on youth or Spanish-speaking populations, so the investigators will obtain feedback on the assessment from these groups.

Aim 2: Evaluate the effectiveness of a youth-led HTN education digital badge intervention on the primary outcome of mean systolic BP and diastolic BP change in adults with uncontrolled HTN at 2-months post-intervention compared to the control group (for participants recruited from the ED). Additionally, evaluate change in HTN knowledge and youth self-efficacy.

Aim 3: Evaluate the implementation process of the youth-led HTN education digital badge by collecting qualitative and quantitative data on acceptability, feasibility, and fidelity of the intervention by participants.

ELIGIBILITY:
Inclusion Criteria:

* Aim 1: Participants will be youth (15-18 years) and adults (18+ years old) with self-reported HTN diagnosis.
* Aim 1a: Participants will be youth (15-18 years) and Spanish-speaking adults (18+ years old) with self-reported HTN diagnosis.
* Aim 2: ED cohort: Eligible adult participants will be 18+ year old ED patients with a history of HTN and two high BP (≥ 130/80 mmHg) readings during their ED visit who know a 14-24 year old. The eligible youth participants (14-24- year-old) must have access to the internet or data plan and a smart phone or computer.

School cohort: Youth Eligibility: Any interested student at New Brunswick Health Sciences Technology High School.

Adult Eligibility: Adult (18+) (preference for adult who has been diagnosed with hypertension) with an existing relationship with the youth where it would be feasible to complete an online module together 1 hour per week for 6 weeks. Fluency in English or Spanish (youth must be able to speak fluent language).

* Aim 3: Everyone who consented to the RCT will be asked to complete a questionnaire, regardless of whether they completed the digital badge. Interested participants from the intervention arm will be recruited for the in-depth interviews.

Exclusion Criteria:

* Aim 1: Age <15 years, inability to speak fluently in English or Spanish
* Aim 1a: Age <15 years, inability to speak fluently in English or Spanish
* Aims 2 and 3: ED cohort: Age <14 years, inability to speak fluently in English or Spanish, no access to the internet or a data plan and a smart phone or computer.

School cohort: People who cannot take part in the study are people who are not able to speak fluently in English or Spanish (youth and adult must be able to speak the same language), and youth with no access to the internet or a data plan and a smart phone or computer.

* Aim 3 (interviews): Participants from the control arm will not be eligible for the in-depth interviews.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-10-31 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to recruitment challenges for the ED cohort, Aim 2 of the study was changed from recruitment in the ED to recruitment in a school. Hence, we only have data for the school cohort. Additionally, the number of participants represents both members of each dyad (adults and youth) combined.
Groups:
- Aim 2 School Cohort: The intervention is a youth-led HTN education digital intervention, which will be comprised of a 6-week playlist of one module per week comprising the playlist. Youth will learn from the module and will teach the adult in their dyad about hypertension education in each week's themed module.
  Youth-Led Hypertension Education Digital Intervention: The intervention is a youth-led HTN education digital intervention, which will be comprised of a 6-week playlist of one module per week comprising the playlist. Youth will learn from the module and will teach the adult in their dyad about hypertension education in each week's themed module.
  The number of people listed here are adults and youth combined (total number of people, not dyads).
- Aim 1 Participants: Qualitative interviews and focus groups to develop the intervention.
- Aim 2 ED Cohort: Participants recruited in the ED for Aim 2 of study. Enrollment was very low with less engagement and no dyads completed the intervention, so shifted to recruitment in the school.
Period: Overall Study
Arm/Group | Aim 2 School Cohort | Aim 1 Participants | Aim 2 ED Cohort
Started (19 adults and 19 youth) | 38 | 22 (12 youth and 10 adults) | 4 (2 adults and 2 youth)
Completed (15 adults and 15 youth) | 30 | 22 (12 youth and 10 adults) | 0
Not Completed | 8 | 0 | 4
Not completed — Withdrawal by Subject | 4 | 0 | 2
Not completed — Lost to Follow-up | 4 | 0 | 2

BASELINE CHARACTERISTICS:
Population: 34 participants enrolled in Aim 2: School, 22 participants enrolled in Aim 1, 4 participants enrolled in Aim 2: ED Cohort (none completed the study from the ED cohort).
Groups:
- Aim 2: School Cohort: The intervention is a youth-led HTN education digital intervention, which will be comprised of a 6-week playlist of one module per week comprising the playlist. Youth will learn from the module and will teach the adult in their dyad about hypertension education in each week's themed module.
  Youth-Led Hypertension Education Digital Intervention: The intervention is a youth-led HTN education digital intervention, which will be comprised of a 6-week playlist of one module per week comprising the playlist. Youth will learn from the module and will teach the adult in their dyad about hypertension education in each week's themed module.
- Aim 1 Participants: To develop the youth-led HTN digital intervention, we conducted a formative study to determine acceptable and easily comprehensible ways to present hypertension information to adults with hypertension and optimal ways to engage youth to support adults on how to achieve better hypertension control. After creating an intervention prototype with 6 weekly self-guided hypertension online modules, we recruited 12 youth (adolescents, aged 15-18 years) for 3 focus groups and 10 adult ED patients with hypertension for individual online interviews to garner feedback on the prototype. After completing a brief questionnaire, participants were asked about experiences with hypertension, preferences for a hypertension education intervention, and acceptability, feasibility, obstacles, and solutions for intervention implementation with youth and adults.
- Aim 2: ED Cohort: We found little success recruiting participants through the emergency department. No participants completed the study and we shifted to recruitment through a local high school (see Aim 2: School Cohort).
- Total: Total of all reporting groups
Arm/Group | Aim 2: School Cohort | Aim 1 Participants | Aim 2: ED Cohort | Total
Number analyzed (Participants) | 34 | 22 | 4 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: This is a dyad study of adult-youth dyads so adult and youth participants are separated.
  years
    Youth: number analyzed (Participants) | 17 | 12 | 2 | 31
    Youth | 15.5 (1.1) | 15.9 (0.8) | 20.0 (4.2) | 15.9 (1.6)
    Adults: number analyzed (Participants) | 17 | 10 | 2 | 29
    Adults | 43.3 (4.7) | 49.8 (17.0) | 61.5 (20.5) | 47.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: This is a dyad study of adult-youth dyads so adult and youth participants are separated.
  Participants
    Youth: number analyzed (Participants) | 17 | 12 | 2 | 31
    Youth: Female | 17 | 7 | 1 | 25
    Youth: Male | 0 | 5 | 1 | 6
    Adults: number analyzed (Participants) | 17 | 10 | 2 | 29
    Adults: Female | 13 | 4 | 2 | 19
    Adults: Male | 4 | 6 | 0 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: This is a dyad study of adult-youth dyads so adult and youth participants are separated.
  Participants
    Youth: number analyzed (Participants) | 17 | 12 | 2 | 31
    Youth: American Indian or Alaska Native | 2 | 0 | 0 | 2
    Youth: Asian | 1 | 1 | 1 | 3
    Youth: Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 2
    Youth: Black or African American | 0 | 1 | 1 | 2
    Youth: White | 8 | 4 | 0 | 12
    Youth: More than one race | 1 | 0 | 0 | 1
    Youth: Unknown or Not Reported | 3 | 6 | 0 | 9
    Adults: number analyzed (Participants) | 17 | 10 | 2 | 29
    Adults: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Adults: Asian | 1 | 4 | 1 | 6
    Adults: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Adults: Black or African American | 0 | 1 | 1 | 2
    Adults: White | 4 | 4 | 0 | 8
    Adults: More than one race | 1 | 1 | 0 | 2
    Adults: Unknown or Not Reported | 11 | 0 | 0 | 11
HTN Knowledge [Mean (Standard Deviation); unit: questions correct out of 21 total] — Population: Aim 2: 17 youth and 17 adults for school cohort and 2 youth and 2 adults for ED cohort.
  This variable was not collected for Aim 1 participants.
  questions correct out of 21 total
    Youth: number analyzed (Participants) | 17 | 0 | 2 | 19
    Youth | 13.0 (3.2) |  | 15 (2.8) | 13.2 (3.2)
    Adults: number analyzed (Participants) | 17 | 0 | 2 | 19
    Adults | 12.3 (4.0) |  | 14 (7.1) | 12.5 (4.3)
Youth- Confidence in Managing High Blood Pressure [Mean (Standard Deviation); unit: units on a scale] — Population: Only measured in youth.
  This variable was not collected for Aim 1 participants.
  units on a scale
    Teach an adult how to lower their high BP.: number analyzed (Participants) | 17 | 0 | 2 | 19
    Teach an adult how to lower their high BP. | 5.6 (3.2) |  | 8 (2.8) | 5.9 (3.2)
    Encourage an adult to lower their high BP.: number analyzed (Participants) | 17 | 0 | 2 | 19
    Encourage an adult to lower their high BP. | 6.9 (2.9) |  | 8 (2.8) | 7.0 (2.9)
    Help an adult lower their BP.: number analyzed (Participants) | 17 | 0 | 2 | 19
    Help an adult lower their BP. | 6.2 (3.4) |  | 8 (2.8) | 6.4 (3.3)
Adult- Blood Pressure Self-Care Scale [Mean (Standard Deviation); unit: units on a scale] — Population: Only measured in adults.
  This variable was not collected for Aim 1 participants.
  units on a scale
    number analyzed (Participants) | 17 | 0 | 2 | 19
    (all) | 3.8 (1.0) |  | 4.6 (0.4) | 3.9 (0.9)
Adult Self-Efficacy to Manage Hypertension Scale [Mean (Standard Deviation); unit: units on a scale] — Population: Only for adults with diagnosed hypertension.
  This variable was not collected for Aim 1 participants.
  units on a scale
    number analyzed (Participants) | 4 | 0 | 2 | 6
    (all) | 6.2 (3.1) |  | 5.8 (4.0) | 6.1 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: School Cohort: Hypertension Knowledge (Youth and Adult)
Description: Using 21-question assessment adapted from Williams et al.'s 1998 hypertension knowledge tool. Results reported are the mean number of questions correct out of 21.
Time Frame: At end of 6-week intervention, and 1 month post-6-week intervention
Population: High Blood Pressure Knowledge (# correct responses), Mean (SD), [95% CI]
Measure: Mean (Standard Deviation); unit: number of questions correct out of 21
Groups:
- Youth; Adults: The intervention is a youth-led HTN education digital intervention, which will be comprised of a 6-week playlist of one module per week comprising the playlist. Youth will learn from the module and will teach the adult in their dyad about hypertension education in each week's themed module.
  Youth-Led Hypertension Education Digital Intervention: The intervention is a youth-led HTN education digital intervention, which will be comprised of a 6-week playlist of one module per week comprising the playlist. Youth will learn from the module and will teach the adult in their dyad about hypertension education in each week's themed module.
Arm/Group | Youth | Adults
Number analyzed (Participants) | 13 | 14
number of questions correct out of 21
  At end of 6-week intervention | 17.5 (1.5) | 17.6 (1.7)
  1 month post-6-week intervention | 17.9 (2.7) | 17.8 (2.4)
Statistical Analysis 1: Comparison: Youth; Comparison of effect size: baseline to post-intervention (d1); Test type: Other — Effect size (Cohen's d); Cohen's d = 1.337 — d1 is mean change from baseline to follow-up divided by the standard deviation of the outcome at baseline to provide an effect size that might approximate one found in a randomized clinical trial if the placebo group saw no change from baseline
Statistical Analysis 2: Comparison: Youth; Comparison of effect size: baseline to post-intervention (d2); Test type: Other — Effect size (Cohen's d); Cohen's d = 1.337 — d2 is mean change from baseline to follow-up divided by the standard deviation of the change from baseline to follow-up, to provide an effect size that would be useful for planning similar before-after studies
Statistical Analysis 3: Comparison: Youth; Comparison of effect size: baseline to 1-month post-intervention (d1); Test type: Other — Effect size (Cohen's d); Cohen's d = 1.300 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Youth; Comparison of effect size: baseline to 1-month post-intervention (d2); Test type: Other — Effect size (Cohen's d); Cohen's d = 1.159 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Adults; Comparison of effect size: baseline to post-intervention (d1); Test type: Other — Effect size (Cohen's d); Cohen's d = 1.065 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Adults; Comparison of effect size: baseline to post-intervention (d2); Test type: Other — Effect size (Cohen's d); Cohen's d = 1.084 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Adults; Comparison of effect size: baseline to 1-month post-intervention (d1); Test type: Other — Effect size (Cohen's d); Cohen's d = 1.316 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Adults; Comparison of effect size: baseline to 1-month post-intervention (d2); Test type: Other — Effect size (Cohen's d); Cohen's d = 1.048 — [estimate comment as in outcome 1, analysis 2]

2. Secondary Outcome: ED Cohort: Hypertension Knowledge (Youth and Adult)
Description: Using assessment adapted from Williams et al.'s 1998 hypertension knowledge tool
Time Frame: Baseline and 1 week and 2 months post-intervention completion
Population: Due to recruitment challenges for the ED cohort, the study was changed from recruitment in the ED to recruitment in a school. Hence, we only have data for the school cohort.
  No participants enrolled in the ED cohort completed the study (1 dyad- 1 adult and 1 youth were lost to follow-up and 1 dyad- 1 adult and 1 youth discontinued the intervention). No outcome data were collected from the ED cohort.
Arm/Group | Intervention Arm
Number analyzed (Participants) | 0

3. Secondary Outcome: ED Cohort: Youth Self-efficacy
Description: Using a 3-item investigator-created assessment tool on confidence in managing high blood pressure
Time Frame: Baseline and 1 week and 2 months post-intervention completion
Population: as for outcome 2
Arm/Group | Intervention Arm
Number analyzed (Participants) | 0

4. Secondary Outcome: School Cohort: Youth Self-efficacy
Description: To measure youth confidence helping an adult manage hypertension, investigators created a 3-item assessment from 1 (not at all confident) to 10 (totally confident), on confidence to 1) teach, 2) encourage, and 3) help an adult lower their BP. The outcome measure represents the mean for each of the three items.
Time Frame: At end of 6-week intervention and 1 month post-6-week intervention
Population: Participants completed the assessment at post-intervention and 1-month post-intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Youth- Post-Intervention; Youth- 1-Month Post-Intervention: The intervention is a youth-led HTN education digital intervention, which will be comprised of a 6-week playlist of one module per week comprising the playlist. Youth will learn from the module and will teach the adult in their dyad about hypertension education in each week's themed module.
  Youth-Led Hypertension Education Digital Intervention: The intervention is a youth-led HTN education digital intervention, which will be comprised of a 6-week playlist of one module per week comprising the playlist. Youth will learn from the module and will teach the adult in their dyad about hypertension education in each week's themed module.
Arm/Group | Youth- Post-Intervention | Youth- 1-Month Post-Intervention
Number analyzed (Participants) | 13 | 13
score on a scale
  Teach an adult how to lower their BP. | 8.2 (1.3) | 8.7 (1.4)
  Encourage an adult to lower their high BP. | 8.9 (1.0) | 9.0 (1.2)
  Help an adult lower their BP. | 8.8 (1.6) | 9.0 (1.3)
Statistical Analysis 1: Comparison: Youth- Post-Intervention; Comparison of effect size: baseline to post-intervention for the statement: "Teach an adult how to lower their high BP." (d1); Test type: Other — Effect size (Cohen's d); Cohen's d = 0.846 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Youth- Post-Intervention; Comparison of effect size: baseline to post-intervention for the statement: "Teach an adult how to lower their high BP." (d2); Test type: Other — Effect size (Cohen's d); Cohen's d = 0.821 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Youth- 1-Month Post-Intervention; Comparison of effect size: baseline to 1-month post-intervention for the statement: "Teach an adult how to lower their high BP." (d1); Test type: Other — Effect size (Cohen's d); Cohen's d = 0.870 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Youth- 1-Month Post-Intervention; Comparison of effect size: baseline to 1-month post-intervention for the statement: "Teach an adult how to lower their high BP." (d2); Test type: Other — Effect size (Cohen's d); Cohen's d = 0.782 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Youth- Post-Intervention; Comparison of effect size: baseline to post-intervention for the statement: "Encourage an adult to lower their high BP." (d1); Test type: Other — Effect size (Cohen's d); Cohen's d = 0.643 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Youth- Post-Intervention; Comparison of effect size: baseline to post-intervention for the statement: "Encourage an adult to lower their high BP." (d2); Test type: Other — Effect size (Cohen's d); Cohen's d = 0.616 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Youth- 1-Month Post-Intervention; Comparison of effect size: baseline to 1-month post-intervention for the statement: "Encourage an adult to lower their high BP." (d1); Test type: Other — Effect size (Cohen's d); Cohen's d = 0.724 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Youth- 1-Month Post-Intervention; Comparison of effect size: baseline to 1-month post-intervention for the statement: "Encourage an adult to lower their high BP." (d2); Test type: Other — Effect size (Cohen's d); Cohen's d = 0.683 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Youth- Post-Intervention; Comparison of effect size: baseline to post-intervention for the statement: "Help an adult lower their BP." (d1); Test type: Other — Effect size (Cohen's d); Cohen's d = 0.720 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Youth- Post-Intervention; Comparison of effect size: baseline to post-intervention for the statement: "Help an adult lower their BP." (d2); Test type: Other — Effect size (Cohen's d); Cohen's d = 0.667 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Youth- 1-Month Post-Intervention; Comparison of effect size: baseline to 1-month post-intervention for the statement: "Help an adult lower their BP." (d1); Test type: Other — Effect size (Cohen's d); Cohen's d = 0.720 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Youth- 1-Month Post-Intervention; Comparison of effect size: baseline to 1-month post-intervention for the statement: "Help an adult lower their BP." (d2); Test type: Other — Effect size (Cohen's d); Cohen's d = 0.627 — [estimate comment as in outcome 1, analysis 2]

5. Secondary Outcome: ED Cohort: Adult Blood Pressure Self-care
Description: Using the Adult Blood Pressure Self-Care Scale (Warren-Findlow et al.)
Time Frame: Baseline and 1 week and 2 months post-intervention completion
Population: as for outcome 2
Arm/Group | Intervention Arm
Number analyzed (Participants) | 0

6. Secondary Outcome: School Cohort: Adult Blood Pressure Self-care
Description: Mean using the 10-question Adult Blood Pressure Self-Care Scale (Peters & Templin, 2010), which states: "In general, how often are the following statements true about you?" on a scale of 1-Never to 7-Always for self-reported frequency of behaviors (e.g. diet, exercise) that control BP. (e.g.: "I am eating a low-salt diet each day.")
Time Frame: At end of 6-week intervention and 1 month post-6-week intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Adult- Post-Intervention; Adult- 1-Month Post-Intervention: The intervention is a youth-led HTN education digital intervention, which will be comprised of a 6-week playlist of one module per week comprising the playlist. Youth will learn from the module and will teach the adult in their dyad about hypertension education in each week's themed module.
  Youth-Led Hypertension Education Digital Intervention: The intervention is a youth-led HTN education digital intervention, which will be comprised of a 6-week playlist of one module per week comprising the playlist. Youth will learn from the module and will teach the adult in their dyad about hypertension education in each week's themed module.
Arm/Group | Adult- Post-Intervention | Adult- 1-Month Post-Intervention
Number analyzed (Participants) | 12 | 14
score on a scale | 4.9 (1.2) | 5.2 (0.9)
Statistical Analysis 1: Comparison: Adult- Post-Intervention; Comparison of effect size: baseline to post-intervention (d1); Test type: Other — Effect size (Cohen's d); Cohen's d = 1.457 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Adult- Post-Intervention; Comparison of effect size: baseline to post-intervention (d2); Test type: Other — Effect size (Cohen's d); Cohen's d = 1.691 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Adult- 1-Month Post-Intervention; Comparison of effect size: baseline to 1-month post-intervention (d1); Test type: Other — Effect size (Cohen's d); Cohen's d = 1.841 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Adult- 1-Month Post-Intervention; Comparison of effect size: baseline to 1-month post-intervention (d2); Test type: Other — Effect size (Cohen's d); Cohen's d = 1.451 — [estimate comment as in outcome 1, analysis 2]

7. Secondary Outcome: ED Cohort: Adult Self-efficacy to Manage HTN
Description: Using Adult Self-Efficacy to Manage Hypertension Scale (Warren-Findlow et al.)
Time Frame: Baseline and 1 week and 2 months post-intervention completion
Population: as for outcome 2
Arm/Group | Intervention Arm
Number analyzed (Participants) | 0

8. Secondary Outcome: School Cohort: Adult Self-efficacy to Manage HTN
Description: Mean using the 5-question Adult Self-Efficacy to Manage Hypertension Scale (Warren-Findlow et al.) which asks about confidence in managing BP control behaviors on a scale of 1-not at all confident to 10-totally confident.
Time Frame: At end of 6-week intervention and 1 month post-6-week intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult- Post-Intervention | Adult- 1-Month Post-Intervention
Number analyzed (Participants) | 3 | 3
score on a scale | 8.1 (1.7) | 8.5 (1.4)
Statistical Analysis 1: Comparison: Adult- Post-Intervention; Comparison of effect size: baseline to post-intervention (d1); Test type: Other — Effect size (Cohen's d); Cohen's d = 0.763 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Adult- Post-Intervention; Comparison of effect size: baseline to post-intervention (d2); Test type: Other — Effect size (Cohen's d); Cohen's d = 1.266 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Adult- 1-Month Post-Intervention; Comparison of effect size: baseline to 1-month post-intervention (d1); Test type: Other — Effect size (Cohen's d); Cohen's d = 0.894 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Adult- 1-Month Post-Intervention; Comparison of effect size: baseline to 1-month post-intervention (d2); Test type: Other — Effect size (Cohen's d); Cohen's d = 1.149 — [estimate comment as in outcome 1, analysis 2]

9. Other Pre Specified Outcome: For ED Cohort: Blood Pressure Change
Description: Change in systolic and diastolic adult blood pressure (in mm Hg)
Time Frame: Baseline to 1 week and 2 months post-intervention completion
Population: Due to recruitment challenges for the ED cohort, the study was changed from recruitment in the ED to recruitment in a school. Hence, we only have data for the school cohort. No outcome data were collected from the ED cohort.
Arm/Group | Intervention Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: Includes adverse events for both adult and youth participants. (No adverse events transpired.)
Arm/Group | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/87/NCT05029687/Prot_SAP_001.pdf
  • Informed Consent Form (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/87/NCT05029687/ICF_002.pdf